CLINICAL TRIAL: NCT00409773
Title: A Multicenter, Randomized, Double-Blind, Parallel Arm, 6-Week Study to Evaluate the Efficacy and Safety of Ezetimibe/Simvastatin Versus Atorvastatin in Patients With Metabolic Syndrome and Hypercholesterolemia at High Risk for Coronary Heart Disease
Brief Title: Ezetimibe/Simvastatin in Patients With Metabolic Syndrome (0653A-107)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-107; 2006_527
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Metabolic Syndrome
MeSH Terms: conditions — Hypercholesterolemia; Metabolic Syndrome | interventions — Ezetimibe, Simvastatin Drug Combination; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Other): Arm 1: drug + comparator + Placebo
  Interventions: Drug: ezetimibe (+) simvastatin; Drug: Comparator: atorvastatin calcium; Drug: Comparator: Placebo (unspecified)
- 2 (Other): Arm 2: drug + comparator + Placebo
  Interventions: Drug: ezetimibe (+) simvastatin; Drug: Comparator: atorvastatin calcium; Drug: Comparator: Placebo (unspecified)
- 3 (Other): Arm 3: drug + comparator + Placebo
  Interventions: Drug: ezetimibe (+) simvastatin; Drug: Comparator: atorvastatin calcium; Drug: Comparator: Placebo (unspecified)
- 4 (Other): Arm 4: drug + comparator + Placebo
  Interventions: Drug: ezetimibe (+) simvastatin; Drug: Comparator: atorvastatin calcium; Drug: Comparator: Placebo (unspecified)
- 5 (Other): Arm 5: drug + comparator + Placebo
  Interventions: Drug: ezetimibe (+) simvastatin; Drug: Comparator: atorvastatin calcium; Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — Ezetimibe (+) simvastatin combination tablet at doses of 10/20 mg or 10/40 mg.
  Other Names: MK0653A; Vytorin®
Drug: Comparator: atorvastatin calcium — Atorvastatin will be supplied in 10mg, 20mg and 40mg tablets.
  Each patient will receive 1 active treatment dose & 2 Placebo doses at randomization according to a predetermined partial blinding schedule to reduce the number of pills from 5 to 3 per patient per day for 6 weeks.
  Other Names: Lipitor ®
Drug: Comparator: Placebo (unspecified) — Atorvastatin Placebo will be supplied in 10mg, 20mg and 40mg tablets.
  ezetimibe/simvastatin Placebo will be supplied in 10/20mg and 10/40mg combination tablets.
  Each patient will receive 1 active treatment dose & 2 Placebo doses at randomization according to a predetermined partial blinding schedule to reduce the number of pills from 5 to 3 per patient per day for 6 weeks.

SUMMARY:
A 6-week clinical trial in patients with metabolic syndrome and hypercholesterolemia at high risk for coronary heart disease to study the effects of ezetimibe/simvastatin and atorvastatin on lipids.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 79 years of age with metabolic syndrome and hypercholesterolemia at high risk for coronary heart disease (CHD) with LDL-C above 70 mg/dL or 100 mg/dL depending on their CHD risk category

Exclusion Criteria:

* A condition which, in the opinion of the investigator, pose a risk to the patient or interfere with participating in the study
* Patient is likely to be greater than 20% noncompliant in taking study medications
* Patients with chronic medical conditions
* Patients with unstable doses of medications
* Pregnant or lactating women, women intending to become pregnant
* Patient is currently receiving prescription therapy with statins or other lipid-altering medications
* Patient with Type 1 or Type 2 diabetes mellitus that is poorly controlled, newly diagnosed, or is taking new or recently adjusted antidiabetic pharmacotherapy (with the exception of +/- 10 units of insulin)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1143 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosen JB, Ballantyne CM, Hsueh WA, Lin J, Shah AK, Lowe RS, Tershakovec AM. Influence of metabolic syndrome factors and insulin resistance on the efficacy of ezetimibe/simvastatin and atorvastatin in patients with metabolic syndrome and atherosclerotic coronary heart disease risk. Lipids Health Dis. 2015 Sep 4;14:103. doi: 10.1186/s12944-015-0075-5. PMID 26336957
- [Derived] Robinson JG, Ballantyne CM, Hsueh W, Rosen J, Lin J, Shah A, Lowe RS, Hanson ME, Tershakovec AM. Achievement of specified low-density lipoprotein cholesterol, non-high-density lipoprotein cholesterol apolipoprotein B, and high-sensitivity C-reactive protein levels with ezetimibe/simvastatin or atorvastatin in metabolic syndrome patients with and without atherosclerotic vascular disease (from the VYMET study). J Clin Lipidol. 2011 Nov-Dec;5(6):474-82. doi: 10.1016/j.jacl.2011.06.004. Epub 2011 Jun 15. PMID 22108151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In 06-Feb-2007:; Last Patient Last Visit 16-Jul-2008
  110 centers worldwide (International, 12 countries)
  Eligible patients include drug-naïve patients or patients rendered naïve with the appropriate prior washout at moderately high or high risk for coronary heart disease.
Pre-assignment Details: Patients were randomized to 1 of 5 treatment groups: ezetimibe/simvastatin combination tablet or atorvastatin alone for 6 weeks stratified according to their baseline risk category stratum (high risk patients with atherosclerotic vascular disease or high risk patients without atherosclerotic vascular disease and moderately high risk patients).
Groups:
- Atorva 10 mg: Atorvastatin 10 mg once daily for 6 weeks
- EZ/Simva 10 mg/20 mg: Ezetimibe (+) simvastatin combination tablet at doses of 10/20 mg
- Atorva 20mg: Atorvastatin 20 mg once daily for 6 weeks
- EZ/Simva 10 mg/40 mg: Ezetimibe (+) simvastatin combination tablet at doses of 10/40 mg
- Atorva 40 mg: Atorvastatin 40 mg once daily for 6 weeks
Period: Overall Study
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Started | 229 | 229 | 229 | 228 | 228
Completed | 220 | 222 | 220 | 216 | 218
Not Completed | 9 | 7 | 9 | 12 | 10
Not completed — Adverse Event | 3 | 4 | 4 | 2 | 6
Not completed — Lost to Follow-up | 6 | 1 | 2 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 2 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1
Not completed — Lack of Eligibility | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg | Total
Number analyzed (Participants) | 229 | 229 | 229 | 228 | 228 | 1143
Age, Continuous [Mean (Full Range); unit: years] | 59.7 [31 to 79] | 59.7 [32 to 78] | 58.2 [33 to 78] | 59.5 [28 to 80] | 58.4 [28 to 79] | 59.1 [28 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 87 | 106 | 104 | 104 | 498
  Male | 132 | 142 | 123 | 124 | 124 | 645
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 17 | 15 | 15 | 18 | 21 | 86
  Black | 13 | 18 | 18 | 12 | 14 | 75
  Other | 27 | 27 | 19 | 27 | 26 | 126
  White | 172 | 169 | 177 | 171 | 167 | 856

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein (LDL-C) at Week 6
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set (FAS): The FAS population includes all randomized patients who took at least 1 dose of study medication and had a baseline (BL) value and at least one post BL value. Post BL measurements up to 3 days following the last dose of double-blind study medication were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 215 | 219 | 215 | 217 | 217
Percent Change | -36.5 [-38.9 to -34.0] | -49.6 [-52.0 to -47.2] | -39.4 [-41.8 to -36.9] | -53.9 [-56.4 to -51.5] | -46.0 [-48.4 to -43.6]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p < 0.001, ANOVA — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -13.1, 95% CI [-16.5 to -9.8], Standard Error of Mean 1.7
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p < 0.001, ANOVA — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -10.2, 95% CI [-13.6 to -6.9], Standard Error of Mean 1.7
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANOVA — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -8.0, 95% CI [-11.3 to -4.6], Standard Error of Mean 1.7

2. Secondary Outcome: Percent Change From Baseline in Total Cholesterol(mg/dL) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 215 | 220 | 216 | 217 | 218
Percent Change | -26.5 [-28.2 to -24.7] | -33.7 [-35.4 to -31.9] | -28.3 [-30.1 to -26.6] | -37.3 [-39.0 to -35.5] | -32.8 [-34.6 to -31.1]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -7.2, 95% CI [-9.6 to -4.8], Standard Error of Mean 1.2
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -5.4, 95% CI [-7.8 to -2.9], Standard Error of Mean 1.2
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -4.4, 95% CI [-6.8 to -2.0], Standard Error of Mean 1.2

3. Secondary Outcome: Percent Change From Baseline in Triglyceride (TG) (mg/dL) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 215 | 220 | 216 | 217 | 218
Percent Change | -21.7 [-25.0 to -17.9] | -23.3 [-26.9 to -18.2] | -27.5 [-30.8 to -22.4] | -29.5 [-32.5 to -25.0] | -30.0 [-34.2 to -26.5]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p = 0.690, Non-parametric ANOVA; ANOVA using normal scores (Tukey method) based on ranks with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -0.9, 95% CI [-5.4 to 3.3]
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p = 0.200, Non-parametric ANOVA; ANOVA using normal scores (Tukey method) based on ranks with terms for treatment and baseline risk stratum; Median Difference (Final Values) = 2.8, 95% CI [-1.6 to 7.1]
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p = 0.480, Non-parametric ANOVA; ANOVA using normal scores (Tukey method) based on ranks with terms for treatment and baseline risk stratum; Median Difference (Final Values) = -0.4, 95% CI [-4.7 to 3.9]

4. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 215 | 219 | 216 | 217 | 217
Percent Change | 3.4 [1.5 to 5.3] | 6.8 [4.9 to 8.7] | 5.6 [3.7 to 7.5] | 8.8 [6.9 to 10.7] | 4.9 [3.0 to 6.8]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p = 0.013, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = 3.4, 95% CI [0.7 to 6.0], Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p = 0.378, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = 1.2, 95% CI [-1.5 to 3.8], Standard Error of Mean 1.3
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p = 0.003, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = 4.0, 95% CI [1.3 to 6.6], Standard Error of Mean 1.3

5. Secondary Outcome: Percent Change From Baseline in Non- High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 215 | 219 | 216 | 217 | 217
Percent Change | -33.5 [-35.6 to -31.3] | -43.8 [-45.9 to -41.7] | -36.5 [-38.6 to -34.4] | -48.3 [-50.5 to -46.2] | -41.4 [-43.6 to -39.3]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -10.3, 95% CI [-13.3 to -7.3], Standard Error of Mean 1.5
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -7.3, 95% CI [-10.2 to -4.3], Standard Error of Mean 1.5
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -6.9, 95% CI [-9.9 to -3.9], Standard Error of Mean 1.5

6. Secondary Outcome: Percent Change From Baseline in Very Low Density Lipoprotein Cholesterol (VLDL-C) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 215 | 217 | 209 | 214 | 216
Percent Change | -17.7 [-21.4 to -14.0] | -18.3 [-22.0 to -14.7] | -21.6 [-25.3 to -17.8] | -23.4 [-27.1 to -19.7] | -22.7 [-26.4 to -19.0]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p = 0.809, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -0.6, 95% CI [-5.7 to 4.5], Standard Error of Mean 2.6
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p = 0.217, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = 3.2, 95% CI [-1.9 to 8.4], Standard Error of Mean 2.6
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p = 0.796, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -0.7, 95% CI [-5.8 to 4.4], Standard Error of Mean 2.6

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein- B (Apo-B) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 211 | 218 | 213 | 214 | 216
Percent Change | -27.9 [-29.9 to -25.9] | -37.2 [-39.2 to -35.3] | -31.9 [-33.9 to -29.9] | -41.1 [-43.1 to -39.1] | -35.8 [-37.8 to -33.8]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -9.4, 95% CI [-12.1 to -6.6], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -5.3, 95% CI [-8.1 to -2.6], Standard Error of Mean 1.4
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -5.3, 95% CI [-8.0 to -2.5], Standard Error of Mean 1.4

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein-A1 (Apo-A1) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 211 | 219 | 213 | 214 | 216
Percent Change | 0.8 [-1.0 to 2.5] | 3.2 [1.5 to 4.9] | 1.0 [-0.7 to 2.7] | 3.0 [1.3 to 4.7] | 1.4 [-0.3 to 3.1]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p = 0.042, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = 2.4, 95% CI [0.1 to 4.8], Standard Error of Mean 1.2
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = 2.2, 95% CI [-0.2 to 4.5], Standard Error of Mean 1.2
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = 1.6, 95% CI [-7.0 to 4.0], Standard Error of Mean 1.2

9. Secondary Outcome: Percent Change From Baseline in Total-Cholesterol: High Density Lipoprotein-Cholesterol (Total-C:HDL- C) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 215 | 219 | 216 | 217 | 217
Percent Change | -28.1 [-30.1 to -26.0] | -36.9 [-38.9 to -34.8] | -31.5 [-33.6 to -29.5] | -41.2 [-43.2 to -39.1] | -35.3 [-37.3 to -33.2]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -8.8, 95% CI [-11.6 to -6.0], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -5.3, 95% CI [-8.2 to -2.5], Standard Error of Mean 1.4
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -5.9, 95% CI [-8.7 to -3.1], Standard Error of Mean 1.4

10. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol: High Density Lipoprotein Cholesterol (LDL-C: HDL-C) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 215 | 219 | 215 | 217 | 217
Percent Change | -37.8 [-40.3 to -35.2] | -51.8 [-54.3 to -49.3] | -42.1 [-44.7 to -39.6] | -56.6 [-59.2 to -54.1] | -48.2 [-50.7 to -45.6]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -14.0, 95% CI [-17.6 to -10.5], Standard Error of Mean 1.8
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -9.7, 95% CI [-13.2 to -6.1], Standard Error of Mean 1.8
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -8.5, 95% CI [-12.0 to -4.9], Standard Error of Mean 1.8

11. Secondary Outcome: Percent Change From Baseline in Apolipoprotein-B: Apolipoprotein-A1 (Apo-B:Apo-A1) at Week 6
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 211 | 218 | 213 | 214 | 216
Percent Change | -27.4 [-29.6 to -25.2] | -38.4 [-40.6 to -36.2] | -32.0 [-34.2 to -29.8] | -41.9 [-44.1 to -39.7] | -36.2 [-38.4 to -34.0]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -11.0, 95% CI [-14.0 to -8.0], Standard Error of Mean 1.5
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -6.4, 95% CI [-9.4 to -3.3], Standard Error of Mean 1.5
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -5.7, 95% CI [-8.7 to -2.7], Standard Error of Mean 1.5

12. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol: High Density Lipoprotein Cholesterol (Non-HDL-C:HDL-C) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 215 | 219 | 216 | 217 | 217
Percent Change | -34.7 [-37.2 to -32.2] | -46.2 [-48.6 to -43.7] | -39.2 [-41.7 to -36.7] | -51.2 [-53.7 to -48.7] | -43.5 [-46.0 to -41.0]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -11.5, 95% CI [-15.0 to -8.1], Standard Error of Mean 1.8
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -7.0, 95% CI [-10.4 to -3.6], Standard Error of Mean 1.8
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with terms for treatment and baseline risk stratum; Mean Difference (Final Values) = -7.7, 95% CI [-11.2 to -4.3], Standard Error of Mean 1.8

13. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 6 in Patients With Atherosclerotic Vascular Disease (AVD)
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 64 | 71 | 59 | 61 | 63
Percent Change | -37.1 [-41.4 to -32.7] | -48.7 [-52.8 to -44.6] | -36.9 [-41.5 to -32.4] | -56.1 [-60.6 to -51.7] | -45.8 [-50.2 to -41.5]

14. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 6 in Patients Without Atherosclerotic Vascular Disease (AVD)
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 151 | 148 | 156 | 156 | 154
Percent Change | -36.3 [-39.1 to -33.5] | -50.1 [-52.9 to -47.2] | -40.3 [-43.1 to -37.6] | -53.2 [-55.9 to -50.4] | -46.1 [-48.9 to -43.3]

15. Secondary Outcome: Percent Change From Baseline in High-Sensitivity C-reactive (Hs-CRP) (mg/dL) at Week 6
Time Frame: Baseline and 6 Weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Number analyzed (Participants) | 216 | 218 | 210 | 216 | 215
Percent Change | -16.8 [-21.7 to -10.6] | -17.2 [-24.1 to -12.5] | -22.4 [-26.1 to -14.6] | -27.6 [-33.3 to -21.4] | -30.0 [-33.3 to -25.0]
Statistical Analysis 1: Comparison: Atorva 10 mg vs EZ/Simva 10 mg/20 mg; Test type: Superiority or Other; p = 0.420, Non-parametric ANOVA; ANOVA using normal scores (Tukey method) based on ranks with terms for treatment and baseline risk stratum; Median Difference (Final Values) = -2.9, 95% CI [-11.0 to 5.0]
Statistical Analysis 2: Comparison: EZ/Simva 10 mg/20 mg vs Atorva 20mg; Test type: Superiority or Other; p = 0.555, Non-parametric ANOVA; ANOVA using normal scores (Tukey method) based on ranks with terms for treatment and baseline risk stratum; Median Difference (Final Values) = -0.9, 95% CI [-9.5 to 7.2]
Statistical Analysis 3: Comparison: EZ/Simva 10 mg/40 mg vs Atorva 40 mg; Test type: Superiority or Other; p = 0.410, Non-parametric ANOVA; ANOVA using normal scores (Tukey method) based on ranks with terms for treatment and baseline risk stratum; Median Difference (Final Values) = 2.3, 95% CI [-5.1 to 9.6]

ADVERSE EVENTS:
Arm/Group | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Serious Adverse Events (participants affected / at risk) | 4 | 0 | 1 | 1 | 4
Other Adverse Events (participants affected / at risk) | 21 | 14 | 22 | 13 | 13
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Acute Myocardial Infarction (Cardiac disorders) | 1/228 | 0/226 | 0/226 | 0/224 | 0/224
Atrial Fibrillation (Cardiac disorders) | 1/228 | 0/226 | 0/226 | 0/224 | 0/224
Atrioventricular Block Second Degree (Cardiac disorders) | 0/228 | 0/226 | 0/226 | 1/224 | 0/224
Sick Sinus Syndrome (Cardiac disorders) | 0/228 | 0/226 | 1/226 | 0/224 | 0/224
Tachyarrhythmia (Cardiac disorders) | 0/228 | 0/226 | 0/226 | 0/224 | 1/224
Cholestasis (Hepatobiliary disorders) | 0/228 | 0/226 | 0/226 | 0/224 | 1/224
Urinary Tract Infection (Infections and infestations) | 0/228 | 0/226 | 1/226 | 0/224 | 0/224
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/226 | 0/226 | 0/224 | 1/224
Cerebrovascular Accident (Nervous system disorders) | 0/228 | 0/226 | 0/226 | 0/224 | 1/224
Headache (Nervous system disorders) | 1/228 | 0/226 | 0/226 | 0/224 | 0/224
Ischaemic Cerebral Infarction (Nervous system disorders) | 1/228 | 0/226 | 0/226 | 0/224 | 0/224
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Atorva 10 mg | EZ/Simva 10 mg/20 mg | Atorva 20mg | EZ/Simva 10 mg/40 mg | Atorva 40 mg
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 7/228 | 6/226 | 7/226 | 4/224 | 2/224
Abdominal Tenderness (Gastrointestinal disorders) | 1/228 | 2/226 | 3/226 | 1/224 | 0/224
Diarrhoea (Gastrointestinal disorders) | 5/228 | 1/226 | 3/226 | 1/224 | 1/224
Nausea (Gastrointestinal disorders) | 1/228 | 3/226 | 1/226 | 2/224 | 1/224
Any General Disorders And Administration Site Conditions (General disorders) | 2/228 | 2/226 | 2/226 | 1/224 | 0/224
Fatigue (General disorders) | 2/228 | 2/226 | 2/226 | 1/224 | 0/224
Any Infections and Infestations (Infections and infestations) | 1/228 | 1/226 | 2/226 | 2/224 | 1/224
Nasopharyngitis (Infections and infestations) | 1/228 | 1/226 | 2/226 | 2/224 | 1/224
Any Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 8/228 | 7/226 | 9/226 | 5/224 | 7/224
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/228 | 1/226 | 1/226 | 2/224 | 1/224
Back Pain (Musculoskeletal and connective tissue disorders) | 0/228 | 2/226 | 0/226 | 3/224 | 2/224
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2/228 | 2/226 | 3/226 | 0/224 | 1/224
Myalgia (Musculoskeletal and connective tissue disorders) | 3/228 | 2/226 | 3/226 | 0/224 | 3/224
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3/228 | 1/226 | 2/226 | 1/224 | 1/224
Any Nervous System Disorders (Nervous system disorders) | 4/228 | 2/226 | 4/226 | 3/224 | 2/224
Dizziness (Nervous system disorders) | 0/228 | 2/226 | 0/226 | 3/224 | 0/224
Headache (Nervous system disorders) | 4/228 | 0/226 | 4/226 | 0/224 | 2/224
Any Vascular Disorders (Vascular disorders) | 2/228 | 0/226 | 0/226 | 0/224 | 2/224
Hypertension (Vascular disorders) | 2/228 | 0/226 | 0/226 | 0/224 | 0/224

LIMITATIONS AND CAVEATS:
15 patients were randomized but not treated. Since these patients were not treated no Adverse Event Data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.